CLINICAL TRIAL: NCT02884323
Title: A Single Centre Open Label Pilot Study Measuring Lower Limb Physiology in Patients With Venous Leg Ulcers Using the Geko™ T-2 or gekoTM Plus [R-2] Neuromuscular Electro Stimulation Device
Brief Title: A Study in Patients With Venous Leg Ulcers and Measuring the Effects of Using Geko™ Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firstkind Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FSK-VLU-002
Record Dates: First submitted 2016-08-17; First posted 2016-08-31 (Estimated); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- geko device arm (Experimental)
  Interventions: Device: geko™ device

INTERVENTIONS:
Device: geko™ device — The geko™ (T-2 and R-2) devices are small disposable, internally powered, neuromuscular stimulators that are applied externally to the leg.

SUMMARY:
This is a single centre open label study measuring lower limb physiology in patients with venous leg ulcers at the University Hospital of South Manchester.

Ambulatory venous pressure, venous transit times, wound bed tissue oxygenation and changes in microcirculation will be measured at baseline after the gekoTM device is activated. Ambulatory venous pressure and venous transit times will be performed whilst the participant is standing, sitting and supine

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Intact healthy skin at the site of device application
3. Able to understand the Patient Information Sheet
4. Willing and able to give informed consent
5. Willing and able to follow the requirements of the protocol
6. Subjects who had a chronic venous leg ulcer (i.e. CEAP classification of C6 1) greater than 1 cm2 and less than 10 cm in maximum diameter,
7. ABPI of ≥0.8
8. Patient treated with 4 layer compression bandaging

Exclusion Criteria:

1. Wound infection either acute or chronic
2. History of significant haematological disorders or DVT with the preceding six months
3. Pregnant
4. Pacemakers or implantable defibrillators
5. Use of any other neuro-modulation device
6. Current use of TENS in pelvic region, back or legs
7. Use of investigational drug or device within the past 4 weeks that may interfere with this study
8. Recent surgery that may affect the study (such as abdominopelvic, or lower limb) in the opinion of the investigator.
9. Recent trauma to the lower limbs
10. Size of leg incompatible with the geko™ device.
11. Obesity (BMI > 34)
12. Any medication deemed to be significant by the Investigator
13. Subjects who had an index venous leg ulcer greater in maximum diameter than 10cm in any one dimension, or less than 2cm.
14. Diabetes
15. Clinical evidence of peripheral arterial disease (i.e signs or symptoms, in the opinion of the researcher)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
The acute effect of the geko™ device on ambulatory venous pressure in patients with venous leg ulcers will be evaluated when sitting, standing or supine | 2 hours
  using Lectromed Multitrace II venous pressure recording system, this will measure Ambulatory venous pressure which will show any influence, if any, gekoTM has on AVP.

SECONDARY OUTCOMES:
The acute effect of the geko™ device on lower leg venous transit times | 2 hours
  Using an ultrasound contrast agent to detect venous flow using Ultrasound imaging. Ultrasound images will be produced and a comparison of results between baseline and using geko™ device will be assessed.
The acute effect of the geko™ device on wound tissue oxygen levels | 2 hours
  The patient will have multipsectral images taken of the ulcer using a fixed camera. The outcome measures (proportions of deoxy- and oxyhaemoglobin) will be displayed on an attached PC.
The effect of the geko™ device on lower leg microcirculation | 2 hours
  Laser Speckle contrast imaging will be applied to record images at baseline and with geko™ device
Adverse events assessments | 2 hours
  Patients will be monitored for adverse events throughout the duration of the study. Adverse events may be spontaneously reported by the subject, observed by the study personnel.
  Serious Adverse Events will be reported to the Sponsor, the National Research Ethics Service (NRES) recognised Research Ethics Committee.

CONTACTS AND LOCATIONS:
Overall Officials: Charles McCollum, Principal Investigator — UHSM
Locations (1):
- The University of Manchester Academic Surgery Unit 2nd Floor, ERC University Hospital of South Manchester M23 9LT, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes